CLINICAL TRIAL: NCT06437496
Title: 68Ga-AAZTA-093 PET/CT: First-in-human Study in Patients With Prostate Cancer
Brief Title: 68Ga-AAZTA-093 PET/CT: First-in-human Study
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FirstAHFujian-68Ga-AAZTA-093
Record Dates: First submitted 2024-05-27; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Malignant Neoplasm of Prostate
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 68Ga-AAZTA-093 PET/ CT (Experimental): Drug: 68Ga-AAZTA-093 Intravenous injection of one dosage of 111-148 MBq (3-4 mCi) 68Ga-AAZTA-093. Tracer doses of 68Ga-AAZTA-093 will be used to image lesions of prostate cancer by PET/CT.
  Interventions: Drug: 68Ga-AAZTA-093
- 68Ga-PSMA-11/68Ga-PSMA-617 PET/ CT (Experimental): Drug: 68Ga-PSMA-11/68Ga-PSMA-617 Intravenous injection of one dosage of 111-148 MBq (3-4 mCi) 68Ga-PSMA-11/68Ga-PSMA-617. Tracer doses of 68Ga-PSMA-11/68Ga-PSMA-617 will be used to image lesions of prostate cancer by PET/CT.
  Interventions: Drug: 68Ga-PSMA-11//68Ga-PSMA-617

INTERVENTIONS:
Drug: 68Ga-AAZTA-093 — Intravenous injection of one dosage of 111-148 MBq (3-4 mCi) 68Ga-AAZTA-093. Tracer doses of 68Ga-AAZTA-093 will be used to image lesions of prostate cancer by PET/CT.
  Arms: 68Ga-AAZTA-093 PET/ CT
Drug: 68Ga-PSMA-11//68Ga-PSMA-617 — Intravenous injection of one dosage of 111-148 MBq (3-4 mCi) 68Ga-PSMA-11//68Ga-PSMA-617. Tracer doses of 68Ga-PSMA-11/68Ga-PSMA-617 will be used to image lesions of prostate cancer by PET/CT.
  Arms: 68Ga-PSMA-11/68Ga-PSMA-617 PET/ CT

SUMMARY:
68Ga-AAZTA-093 is a novel radiotracer targeting prostate-specific membrane antigen (PSMA). In this study, we observed the safety, biodistribution, radiation dosimetry and diagnostic value of 68Ga-AAZTA-093 PET/CT in patients with prostate cancer.

DETAILED DESCRIPTION:
Prostate cancer (PCa) is one of the most common malignancies worldwide in men. Prostate specific membrane antigen (PSMA), as known as folate hydrolase I or glutamate carboxypeptidase II, is overexpressed on the cells of prostatic adenocarcinoma. Various low molecular weight radiopharmaceuticals targeting PSMA such as PSMA-11, PSMA-617 for 68Ga- or 177Lu- labeling have been developed. 68Ga-AAZTA-093, a novel radiopharmaceutical targeting PSMA, with the urea fragment of a conjugate that employs the AAZTA chelator for labeling with 68Ga(III). This pilot study was prospectively designed to evaluate the safety, biodistribution, radiation dosimetry and diagnostic value of 68Ga-AAZTA-093 PET/CT and compared with 68Ga-PSMA-11 and 68Ga-PSMA-617 PET/CT in the same group of prostate cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* confirmed treated or untreated prostate cancer patients;
* 68Ga-AAZTA-093 and 68Ga-PSMA-11/68Ga-PSMA-617 PET/CT within 1 week;
* signed written consent.

Exclusion Criteria:

* known allergy against PSMA;
* any medical condition that in the opinion of the investigator may significantly interfere with study compliance.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation | Within 7 days following PET/CT
  The safety will be assessed by the number and percentage of patients with adverse events; Adverse events were categorized using the Common Toxicity Criteria for Adverse Events 5.0.

SECONDARY OUTCOMES:
Dosimetry data | through study completion, an average of 3 months
  Calculate the absorbed dose of 68Ga-AAZTA-093 in normal organs.

OTHER OUTCOMES:
Diagnostic value | through study completion, an average of 3 months
  Sensitivity and Specificity of 68Ga-AAZTA-093 for prostate cancer in comparison with 68Ga-PSMA-11/68Ga-PSMA-617 PET/CT.
SUV of tumors | through study completion, an average of 3 months
  Compare the SUV of tumors between 68Ga-AAZTA-093 PET/CT and 68Ga-PSMA-11/68Ga-PSMA-617 PET/CT.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China